CLINICAL TRIAL: NCT02742545
Title: Impact of MayoExpertAdvisor (MEA) on Provider Adherence to Guideline Recommended Treatment for Hyperlipidemia, Atrial Fibrillation, and Heart Failure
Brief Title: Impact of MayoExpertAdvisor on Provider Adherence
Acronym: MEA Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Paul M. McKie, M.D., M.D., Cardiology, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-008444
Record Dates: First submitted 2016-04-11; First posted 2016-04-19 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Hyperlipidemia; Atrial Fibrillation; Heart Failure
MeSH Terms: conditions — Hyperlipidemias; Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MayoExpertAdvisor (Experimental): Clinicians in care teams assigned to the intervention arm will have access to MayoExpertAdvisor (MEA) in the electronic medical record (EMR). MEA will provide patient-specific knowledge and treatment suggestions for patients with hyperlipidemia, atrial fibrillation, and/or heart failure via a clickable tab in the Mayo Clinic EMR.
  Interventions: Behavioral: MayoExpertAdvisor
- Usual Care (No Intervention): Clinicians in care teams assigned to the standard of care arm will continue to provide up-to-date, patient-specific guideline-based treatment recommendations as is the standard of care at Mayo Clinic.

INTERVENTIONS:
Behavioral: MayoExpertAdvisor — Access to MayoExpertAdvisor (MEA) in the electronic medical record (EMR). MEA will provide patient-specific knowledge and treatment suggestions for patients with hyperlipidemia, atrial fibrillation, and/or heart failure via a clickable tab in the Mayo Clinic EMR.
  Arms: MayoExpertAdvisor

SUMMARY:
This study evaluates the efficacy of MayoExpertAdvisor (MEA), a knowledge delivery tool, to improve adherence to best practices for patients with hyperlipidemia, atrial fibrillation and heart failure. Half of the clinicians will receive MEA, while the other half will not receive MEA.

The investigators hypothesize care teams with access to MEA will act upon recommendations at a higher rate than those care teams in the standard of care arm without access to MEA.

DETAILED DESCRIPTION:
MEA is designed to increase adherence to consensus national guidelines and quality measures which are the standard of care for hyperlipidemia, atrial fibrillation, and heart failure. These diseases were selected based on national data which suggest there is less than optimal adherence to standard of care therapy and this non-adherence is associated with adverse cardiovascular outcomes.

There are 29 care teams in the Employee and Community Health (ECH) practice. Care teams are comprised of 4-8 clinicians who provide primary care to between 3,000 and 8000 patients. 8 care teams are resident/fellow led and will be excluded from the study. The remaining 21 care teams in the ECH practice will be stratified by clinic location and provider specialty (Internal Medicine, Family Medicine). 20 care teams will then be cluster-randomized to either the intervention arm or standard of care arm.

Prior to randomization, clinicians in both arms will receive the same educational module to the current guidelines for management of the atrial fibrillation, heart failure and hyperlipidemia. Clinicians in the intervention arm will receive training by the research team on the use of MEA. This training will clearly inform clinicians that they are always to use their best clinical judgment.

ELIGIBILITY:
Clinician Inclusion Criteria:

* Physicians
* Assistants
* Nurse Practitioners

Clinician Exclusion Criteria:

* Clinicians providing care to nursing home patients
* Pediatricians
* Residents and fellows

Patient Record Inclusion Criteria:

* Diagnosis of hyperlipidemia, atrial fibrillation, and/or heart failure

Patient Record Exclusion Criteria:

* Unscheduled visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2248 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Percentage of pre-visit recommendations for hyperlipidemia acted upon by providers | Baseline to 6 months
Percentage of pre-visit recommendations for atrial fibrillation acted upon by providers | Baseline to 6 months
Percentage of pre-visit recommendations for heart failure acted upon by providers | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul M McKie, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Patient identifiers will be removed from the data prior to submission to the researchers.

REFERENCES:
- [Derived] McKie PM, Kor DJ, Cook DA, Kessler ME, Carter RE, Wilson PM, Pencille LJ, Hickey BC, Chaudhry R. Computerized Advisory Decision Support for Cardiovascular Diseases in Primary Care: A Cluster Randomized Trial. Am J Med. 2020 Jun;133(6):750-756.e2. doi: 10.1016/j.amjmed.2019.10.039. Epub 2019 Dec 18. PMID 31862329
- [Derived] Kessler ME, Carter RE, Cook DA, Kor DJ, McKie PM, Pencille LJ, Scheitel MR, Chaudhry R. Impact of electronic clinical decision support on adherence to guideline-recommended treatment for hyperlipidaemia, atrial fibrillation and heart failure: protocol for a cluster randomised trial. BMJ Open. 2017 Dec 4;7(12):e019087. doi: 10.1136/bmjopen-2017-019087. PMID 29208620
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials